CLINICAL TRIAL: NCT03975218
Title: Involvement of the Physician in Primary Prevention and Pre-hospital Management of Stroke
Acronym: PREVENTION AVC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PREVENTION AVC
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stroke: In addition to the usual care, the patient will have to complete a questionnaire analyzing the regularity of his follow-up by a physician.
  Interventions: Other: Patients With Stroke

INTERVENTIONS:
Other: Patients With Stroke — In addition to the usual care, the patient will have to complete a questionnaire analyzing the regularity of his follow-up by a physician.

SUMMARY:
Stroke is a growing disease. It is the first pathology responsible for acquired handicap, the second of dementia and the second cause of death in the world. In France, they are the leading cause of death in women and the third cause in men. Sequelae and disabilities also represent a significant financial cost for health insurance.

The early management of the treatment improves the patient's vital and functional prognosis. The ability of the patient to identify the signs of stroke requiring urgent consultation and proper orientation are therefore crucial for further management.

The most common signs that patients must recognize are muscle weakness or sudden paralysis of an arm, leg or half of the body, asymmetry of the face, tingling, numbness of a hemi-body, speech or understanding, loss of vision of an eye or hemifield, disorder of the coordination of a hemi-body. The variety of clinical pictures complicates primary prevention.

In this context, a 2010-2014 National Stroke Action Plan was undertaken with the aim, among other things, of developing information to prevent stroke and to limit its sequelae. In this plan, the attending physician must improve prevention in high-risk patients and be a link between the city and the hospital for follow-up.

Several questions arise:

* Are patients who are regularly followed by a general practitioner better educated on the signs of stroke / TIA and thus more able to give an appropriate warning?
* What is the profile of patients who have not been affected by the different modes of primary prevention?
* What are the effective means of information and those desired

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient hospitalized in the neurology / neurovascular department within the GHPSJ following a stroke (first episode or recurrence)
* Francophone patient

Exclusion Criteria:

* Patient with previously labeled cognitive impairment
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient unable to answer the questionnaire
* Patient opposing participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in the neurology / neurovascular department within the GHPSJ following a stroke (first episode or recurrence)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Time until patient's care in the hospital after stroke's symptoms | Day 1
  The delay between the observation of signs of stroke and specialized neurovascular management at the hospital will be measured. This measures the impact of physician's prevention on the management of stroke.

SECONDARY OUTCOMES:
Study the different effective means of primary prevention | Day 1
  Patient questionnaire corresponds to open question about physician in primary prevention and pre-hospital management of stroke to which the patient will respond yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Marie BRUANDET, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided